CLINICAL TRIAL: NCT07331714
Title: Comparative Effects of Proprioceptive Neuromuscular Facilitation and Modified Constraint Induced Movement Therapy on Lower Limb Function in Patient With Stroke
Brief Title: Comparative Effects of PNF and mCIMT on Lower Limb Function in Patient With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0294
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: ischemic stroke; stroke rehablitation; stroke; PNF; mCIMT; ROM; Quality of life; Muscle strength; motor function
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF (Experimental): First receive a general preparatory treatment, including hot pack and TENS for 10 minutes to facilitate relaxation, followed by active range of motion exercises as baseline therapy The intervention focused on PNF diagonal patterns, rhythmic initiation, resistance training and dynamic reversals.
  Interventions: Other: PNF
- mCIMT (Experimental): Initially all participants will receive baseline treatment which include general relaxation followed by AROM. Limb will be constraint to 2.5 hours for 5 days a week and therapy time will be 45 minutes focusing on the use of affected limb up to 10 weeks. Side stepping, Ball kicking, Stair climbing, and Knee control on a step.
  Interventions: Other: mCIMT

INTERVENTIONS:
Other: PNF — PNF training was administered for 10 weeks (Time), 5 days per week (Frequency), for 45 minutes per session (Time), using moderate-to-maximal manual resistance (Intensity) with rhythmic initiation, diagonal patterns, dynamic reversals, and resistance training (Type)
  Arms: PNF
Other: mCIMT — mCIMT was administered for 10 weeks (Duration), 5 days per week (Frequency), for 45 minutes per session (Time), involving task-oriented lower limb activities including side stepping, ball kicking, stair climbing, and knee control on a step (Type), performed at moderate functional intensity (Intensity).
  Arms: mCIMT

SUMMARY:
Stroke, which is frequently characterized by weakness, poor balance, and decreased mobility that impede independence in everyday activities, has been identified as a major cause of long-term impairment globally. There have been reports of an increasing number of stroke survivors in Pakistan, however access to proper rehabilitation is sometimes hampered by a lack of resources and awareness. It is thought that improving walking ability, balance, and day-to-day functioning requires the restoration of lower limb function. Modified Constraint-Induced Movement Therapy (mCIMT) and Proprioceptive Neuromuscular Facilitation (PNF) have been found to be successful physiotherapy interventions for improving motor recovery, but there is little comparative data on their impact on lower limb function.

The purpose of this study is to examine the effects of PNF and mCIMT in order to identify whether strategy is better for lower limb rehabilitation after stroke. The findings are expected to give physiotherapists evidence-based recommendations for treatment choices, enabling stroke patients to recover more quickly and become more independent. In the end, community-level advantages are anticipated in the form of less impairment, less caregiver stress, and an overall improvement in the quality of life for stroke victims.

ELIGIBILITY:
Inclusion Criteria:

Patients who are chronic stroke post-stroke or longer will be included. Both males and females are included. Stroke between ages 45 -75 years. Mild to moderate disability assessed using the Modified Rankin Scale (mRS) with a score of 2 to 3.

Pain more than 4 on visual analogue scale in the affected lower limb.

Exclusion Criteria:

Recurring stroke Cognitive impairment (Less than 24 points on Mini Mental Status Examination) Peripheral vascular disease (such as Parkinsonism, epilepsy, multiple sclerosis, or spinal cord injury.

No surgical procedure performed on lower limbs

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
motor function | 10 week
  The Fugl-Meyer Assessment of Lower Extremity (FMA-LE) is a widely used and recommended scale for evaluation of post-stroke motor impairment. The FMA-LE is a reliable tool for assessment of motor impairment both within and between raters early after stroke. The scale can be recommended internationally. A unified international use of FMA-LE would allow comparison of stroke recovery outcomes worldwide and thereby potentially improve the quality of stroke rehabilitation. The scale is recognized as a gold standard and is recommended both for clinical use and research world wide. The scale includes assessment of reflex activity, voluntary movements within and outside of synergies, ability to perform isolated movement, and coordination. This means that the scale is valid for determining level of motor function in people with stroke.The total score of the Fugl-Meyer Assessment for the Lower Extremity (FMA-LE) is 34 points.Each item is scored on a 0-2 scale.
Muscle Strength | 10 week
  The Motricity Index (MI) is an ordinal measure used to assess muscle strength in individuals with post-stroke hemiparesis, originally developed by Demeurisse et al. in 1980. It evaluates three key upper limb movements-pinch grip (PG), elbow flexion (EF), and shoulder abduction (SA)-and three lower limb movements-ankle dorsiflexion (AD), knee extension (KE), and hip flexion (HF), each graded using the Medical Research Council (MRC) 6-point scale and then converted into modified weighted scores. A total score ranging from 0 (complete paresis) to 100 (normal strength) is computed for each limb, and a side score may also be obtained by averaging upper and lower limb totals. Administration time ranges from 5 to 20 minutes depending on the examiner's experience and the severity of impairment. The MI demonstrates excellent inter-rater reliability, strong construct and concurrent validity with established motor impairment scales, and good predictive validity as initial MI scores correlates
range of motion | 10 week
  Goniometer refers to the measurement of angles in particular the measurement of angles created at human joints by the bones of the body. These measurement are obtained by placing the parts of measuring instrument, called a goniometer. Goniometery may be used to determine both a particular joint position and the total amount of motion available at a joint. The data analysis revealed the inter tester reliability and validity were high
stroke specific quality of life | 10 week
  Stroke-specific quality of life (SS-QOL) is a standardized, reliable, and disease-specific questionnaire designed to evaluate quality of life in individuals with stroke. It consists of twelve domains and forty-nine items, each scored on a 5-point Likert scale. The domains include energy, language, mobility, self-care, family roles, social roles, vision, mood, thinking, upper extremity function, and work and productivity. The SS-QOL has been widely validated and is considered an effective tool for assessing functional and psychosocial outcomes in stroke patients.Stroke-Specific Quality of Life (SS-QOL) scale consists of 49 items across 12 domains.Each item is scored on a 5-point Likert scale (1-5). Minimum possible total score is 49 and maximum possible total score is 245.Higher scores indicate better quality of life in stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Riffat Malik, Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Complex Hanjerwal, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bingol H, Gunel MK. Comparing the effects of modified constraint-induced movement therapy and bimanual training in children with hemiplegic cerebral palsy mainstreamed in regular school: A randomized controlled study. Arch Pediatr. 2022 Feb;29(2):105-115. doi: 10.1016/j.arcped.2021.11.017. Epub 2022 Jan 14. PMID 35039189
- [Background] Sharma S, Mehta S. Effectiveness of Lower Limb Proprioceptive Neuromuscular Facilitation on ADL in Stroke.
- [Background] Patni HY. A comparative study on the effects of pelvic PNF exercises and hip extensor strengthening exercises on gait parameters of chronic hemiplegic patients. Int J Physiother Res. 2019;7(4):3150-56.
- [Background] Hussein ZA, Khazraji RTT, Gazi HK. The Efficacy of Strengthening and Stretching by PNF for Foot Drop in Hemiplegia. Iranian Rehabilitation Journal. 2025;23(3):331-8.
- [Background] Chavan NS, Raghuveer R. Lower limb rehabilitation using modified constraint-induced movement therapy and motor relearning program on balance and gait in sub-acute hemiplegic stroke: a comparative study. F1000Res. 2024 Mar 28;12:1098. doi: 10.12688/f1000research.138127.2. eCollection 2023. PMID 39291140
- [Background] Huang S, Zhang Y, Liu P, Chen Y, Gao B, Chen C, Bai Y. Effectiveness of contralaterally controlled functional electrical stimulation vs. neuromuscular electrical stimulation for recovery of lower extremity function in patients with subacute stroke: A randomized controlled trial. Front Neurol. 2022 Dec 8;13:1010975. doi: 10.3389/fneur.2022.1010975. eCollection 2022. PMID 36570446
- [Background] Arif T, Raza T, Saleem Z, Saeed Z, Tariq R, Shahid I. Quality of Life Among Stroke Survivors; A Descriptive Study. Journal Riphah College of Rehabilitation Sciences. 2023;11(03).
- [Background] Hernandez ED, Forero SM, Galeano CP, Barbosa NE, Sunnerhagen KS, Alt Murphy M. Intra- and inter-rater reliability of Fugl-Meyer Assessment of Lower Extremity early after stroke. Braz J Phys Ther. 2021 Nov-Dec;25(6):709-718. doi: 10.1016/j.bjpt.2020.12.002. Epub 2020 Dec 17. PMID 33358073
- [Background] Norkin CC, White DJ. Measurement of joint motion: a guide to goniometry: FA Davis; 2016.
- [Background] Longo D, Doronzio S, Piazzini M, Politi AM, Ciapetti T, Gerli F, Barnabe M, Ciullini F, Castagnoli C, Pellegrini I, Cannobio M, Bardi D, Baccini M, Cecchi F. Development of the Italian version of the Motricity Index and evaluation of its reliability in adults with stroke. J Rehabil Med. 2025 Jan 3;57:jrm40441. doi: 10.2340/jrm.v57.40441. PMID 39749422
- [Background] Lee D, Bae Y. Short-Term Effect of Kinesio Taping of Lower-Leg Proprioceptive Neuromuscular Facilitation Pattern on Gait Parameter and Dynamic Balance in Chronic Stroke with Foot Drop. Healthcare (Basel). 2021 Mar 3;9(3):271. doi: 10.3390/healthcare9030271. PMID 33802448
- [Background] Shahid Z, Dioso RIP. Comparison of Tele-Rehabilitation-Based Training and generic Home-Based Program in Enhancing Balance and Quality of Life in Chronic Stroke Patients: An Experimental Study. 2023.
- [Background] Ceylan CM, Şen Eİ, Karaagac T, Şahbaz T, Yalıman A. Effect of Modified Constraint-Induced Movement Therapy on Upper Extremity Function for Stroke Patients with Right/Left Arm Paresis: A Single-Blind Randomized Controlled Trial. Ahi Evran Medical Journal. 2023;7(2):155-64.
- [Background] Noor S, Bukhari SN, Tariq R, Inam AB. Effect of Modified Constraint Induced Movement Therapy on Improving Hand Function of Stroke Patients. Journal of Islamic International Medical College (JIIMC). 2020;15(4):236-40.
- [Background] Cao M, Li X. Effectiveness of modified constraint-induced movement therapy for upper limb function intervention following stroke: A brief review. Sports Med Health Sci. 2021 Aug 10;3(3):134-137. doi: 10.1016/j.smhs.2021.08.001. eCollection 2021 Sep. PMID 35784520
- [Background] Choi AY, Lim JH, Kim BG. Effects of muscle strength exercise on muscle mass and muscle strength in patients with stroke: a systematic review and meta-analysis. J Exerc Rehabil. 2024 Oct 25;20(5):146-157. doi: 10.12965/jer.2448428.214. eCollection 2024 Oct. PMID 39502116
- [Background] Chaturvedi P. Effects of early proprioceptive neuromuscular facilitation exercises on functional outcome and quality of life in patients with stroke. Age (mean±SD). 2017;61(10.44):55.29-11.07.
- [Background] Abba M, Muhammad A, Badaru U, Abdullahi A. Comparative effect of constraint-induced movement therapy and proprioceptive neuromuscular facilitation on upper limb function of chronic stroke survivors. Physiotherapy Quarterly. 2020;28(1):1-5.
- [Background] Li Y-F. Effectiveness of proprioceptive neuromuscular facilitation techniques in improving balance in poststroke patients: A systematic review. Brain Network and Modulation. 2022;1(1):9-12.
- [Background] Psychouli P, Mamais I, Anastasiou C. An Exploration of the Effectiveness of Different Intensity Protocols of Modified Constraint-Induced Therapy in Stroke: A Systematic Review. Rehabil Res Pract. 2023 Oct 10;2023:6636987. doi: 10.1155/2023/6636987. eCollection 2023. PMID 37854484
- [Background] KALITA SS, SARMA B, HAZARIKA S, DUTTA A. Effect of Proprioceptive Neuromuscular Facilitation Technique on Balance in Stroke Patients: A Narrative Review. Journal of Clinical & Diagnostic Research. 2024;18(6).
- [Background] Umar L, Adegoke B, Dada O. EFFECTS OF MODIFIED CONSTRAINT-INDUCED MOVEMENT THERAPY UPPER AND LOWER LIMBS ON FUNCTIONAL MOBILITY IN STROKE PATIENTS: A RANDOMISED CONTROLLED TRIAL. Journal of Biomedical Investigation. 2024;12(2):94-110.
- [Background] Sethi R, Khalid F, Saghir M, Khan UA, Hanif K. Effects of modified constraint induced movement therapy versus proprioceptive neuromuscular facilitation on upper limb motor function in chronic ischemic stroke patients. Journal Riphah College of Rehabilitation Sciences. 2024;12(2).
- [Background] TM SNK. Comparing the Effect of Proprioceptive Neuromuscular Facilitation (PNF) Exercise and Focused Regimen Program to Assess Balance and Quality of Life for Acute Stroke Rehabilitation. Indian Journal of Physiotherapy & Occupational Therapy. 2024;18.
- [Background] Dioso RIP, Asghar M. Comparison of Effects of Conventional Constrained Induced Movement Therapy Versus Proprioceptive Neuromuscular Facilitation Technique to Improve Functional Motor Skills and Spasticity for Hemiparetic Upper Limb in Sub-Acute Stroke Patients. Insights-Journal of Health and Rehabilitation. 2024;2(2 (Rehab.)):13-8.
- [Background] Candan SA, Livanelioğlu A. Efficacy of modified constraint induced movement therapy for lower extremity in patients with stroke: Strength and quality of life outcomes. Fizyoterapi Rehabilitasyon. 2019;30(1):23-32.
- [Background] Kachhwani N, Qureshi MI, Kovela RK. Effectiveness of proprioceptive neuromuscular facilitation techniques in Improving muscle strength in a patient with hemiplegia. Res Dev. 2022;11:45-7.
- [Background] Srinayanti Y, Widianti W, Andriani D, Firdaus FA, Setiawan H. Range of motion exercise to improve muscle strength among stroke patients: a literature review. International Journal of Nursing and Health Services (IJNHS). 2021;4(3):332-43.
- [Background] Kuriakose D, Xiao Z. Pathophysiology and Treatment of Stroke: Present Status and Future Perspectives. Int J Mol Sci. 2020 Oct 15;21(20):7609. doi: 10.3390/ijms21207609. PMID 33076218
- [Background] Banda KJ, Chu H, Kang XL, Liu D, Pien LC, Jen HJ, Hsiao SS, Chou KR. Prevalence of dysphagia and risk of pneumonia and mortality in acute stroke patients: a meta-analysis. BMC Geriatr. 2022 May 13;22(1):420. doi: 10.1186/s12877-022-02960-5. PMID 35562660
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228
- [Background] Wolfe CD. The impact of stroke. Br Med Bull. 2000;56(2):275-86. doi: 10.1258/0007142001903120. PMID 11092079